CLINICAL TRIAL: NCT03289091
Title: Effects of Two Water-based Aerobic Training Programs on Cardiorespiratory and Neuromuscular Parameters in Elderly Women: a Randomized Controlled Trial
Brief Title: Effects of Two Water-based Aerobic Training Programs in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Stephanie Santana Pinto, Professor in Physical Education School, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WATER
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Elderly Women
Keywords: aerobic training; aquatic exercise; aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- water-based continuous aerobic training (Experimental): Participants who will be randomized for the intervention in the continuous aerobic training group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle. In the first mesocycle (weeks 1-4), participants will carry out three 4-minute series of each exercise whose intensity corresponds to the Rating of Perceived Exertion (RPE) 13. In the second mesocycle (weeks 5-8), participants will perform four 3-minute series of each exercise corresponding to RPE 14. In the third mesocycle, participants will perform six 2-minute series of each exercise at intensity corresponding to RPE 15 from weeks 9-10, whereas intensity corresponding to RPE 16 will be experienced from weeks 11-12.
  Interventions: Behavioral: water-based continuous aerobic training
- water-based interval aerobic training (Experimental): Participants who will be randomized for the intervention in the interval aerobic training group will carry out exercises which associate effort phases, at higher intensity and recovery phases, at lower intensity, with no interval for exercise change. Intensity will be increased every mesocycle. The first mesocycle (weeks 1-4) comprises three 4-minute series of each exercise whose intensity corresponds to the RPE 16 for 2 minutes and RPE 11 for 2 minutes. The second mesocycle (weeks 5-8) includes four 3-minute series of each exercise whose intensity corresponds to the RPE 17 for 1.5 minutes and RPE 11 for 2 minutes. The third mesocycle (weeks 9-12) comprises six 2-minute series of each exercise whose intensity corresponds to the RPE 18 for 1 minute and RPE 11 for 1 minute.
  Interventions: Behavioral: water-based interval aerobic training

INTERVENTIONS:
Behavioral: water-based continuous aerobic training — Participants who will be randomized for the continuous aerobic training group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle. In the first mesocycle (weeks 1-4), participants will carry out three 4-minute series of each exercise whose intensity corresponds to the Rating of Perceived Exertion (RPE) 13. In the second mesocycle (weeks 5-8), participants will perform four 3-minute series of each exercise corresponding to RPE 14. In the third mesocycle, participants will perform six 2-minute series of each exercise at intensity corresponding to RPE 15 from weeks 9-10, whereas intensity corresponding to RPE 16 will be experienced from weeks 11-12.
  Arms: water-based continuous aerobic training
Behavioral: water-based interval aerobic training — Participants who will be randomized for interval aerobic training group will carry out exercises which associate effort phases, at higher intensity and recovery phases, at lower intensity, with no interval for exercise change. Intensity will be increased every mesocycle. The first mesocycle (weeks 1-4) comprises three 4-minute series of each exercise whose intensity corresponds to the RPE 16 for 2 minutes and RPE 11 for 2 minutes. The second mesocycle (weeks 5-8) includes four 3-minute series of each exercise whose intensity corresponds to the RPE 17 for 1.5 minutes and RPE 11 for 2 minutes. The third mesocycle (weeks 9-12) comprises six 2-minute series of each exercise whose intensity corresponds to the RPE 18 for 1 minute and RPE 11 for 1 minute.
  Arms: water-based interval aerobic training

SUMMARY:
The aim of the study is to investigate the effects of two water based aerobic training programs on cardiorespiratory, neuromuscular and quality of life parameters in old women.

Volunteer old women age range: 60-75 years old, will participate to this study, and will randomly divided into two groups: continuous aerobic training group and interval aerobic training group.

Both group subjects will participate in two-week training sessions during 12 weeks. Independent of the group, participants will perform three water-based exercises: stationary running, frontal kick and cross-country skiing. The intensity of aerobic exercise will be based Rating Perceived Exertion (RPE). Along the training, the intensity of aerobic exercise will increase in both groups. Before and after intervention, there will be evaluation of muscle quality, muscle thickness, peak oxygen uptake and oxygen uptake at ventilatory threshold, maximal isometric and dynamic strength of knee extensors, maximal and submaximal isometric eletromiografy (EMG) activity of vastus lateralis and rectus femoris, muscle endurance, performance in functional tests and assessment of the perception of quality of life.

Data will be analyzed by Generalized Estimating Equations (GEE) and Bonferroni's post-hoc test (α=0.05), including both protocol and intention to treat analyses (α=0,05).

DETAILED DESCRIPTION:
Aging is associated with impairment in cardiorespiratory fitness, strength performance and muscle mass decrease, which affects the functional capacity of older adults directly. Consequently carrying out routine activities can be harmed. However regular exercise practice points out as an efficient tool to mitigate factors associated with aging.

Therefore, carrying out water-based exercises has been widely suggested for older adults due to their advantages, such as low impact on lower limbs and lower cardiovascular load.

The aim of the study is to investigate the effects of two water based aerobic training programs on cardiorespiratory, neuromuscular and quality of life parameters in old women.

Volunteer old women age range: 60-75 years old, will participate to this study, and will randomly divided into two groups: continuous aerobic training group and interval aerobic training group.

Both group subjects will participate in two-week training sessions during 12 weeks. Independent of the group, participants will perform three water-based exercises: stationary running, frontal kick and cross-country skiing. The intensity of aerobic exerecise will be based Rating Perceived Exertion (RPE). Along the training, the intensity of aerobic exercise will increase.

Participants who will be randomized for the continuous aerobic training group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle. In the first mesocycle (weeks 1-4), participants will carry out three 4-minute series of each exercise whose intensity corresponds to the Rating of Perceived Exertion (RPE) 13. In the second mesocycle (weeks 5-8), participants will perform four 3-minute series of each exercise corresponding to RPE 14. In the third mesocycle, participants will perform six 2-minute series of each exercise at intensity corresponding to RPE 15 from weeks 9-10, whereas intensity corresponding to RPE 16 will be experienced from weeks 11-12.

Participants who will be randomized for interval aerobic training group will carry out exercises which associate effort phases, at higher intensity and recovery phases, at lower intensity, with no interval for exercise change. Intensity will be increased every mesocycle. The first mesocycle (weeks 1-4) comprises three 4-minute series of each exercise whose intensity corresponds to the RPE 16 for 2 minutes and RPE 11 for 2 minutes. The second mesocycle (weeks 5-8) includes four 3-minute series of each exercise whose intensity corresponds to the RPE 17 for 1.5 minutes and RPE 11 for 2 minutes. The third mesocycle (weeks 9-12) comprises six 2-minute series of each exercise whose intensity corresponds to the RPE 18 for 1 minute and RPE 11 for 1 minute.

Before and after intervention, there will be evaluation of muscle quality, muscle thickness, peak oxygen uptake and oxygen uptake at ventilatory threshold, maximal isometric and dynamic strength of knee extensors, maximal and submaximal isometric eletromiografy (EMG) activity of vastus lateralis and rectus femoris, muscle endurance, performance in functional tests and assessment of the perception of quality of life.

Data will be analyzed by Generalized Estimating Equations (GEE) and Bonferroni's post-hoc test (α=0.05), including both protocol and intention to treat analyses (α=0,05).

ELIGIBILITY:
Inclusion Criteria:

Volunteer elderly women, aged between 60-75 years old who were not participating on any regular training program in the last six months.

Exclusion Criteria:

* Cardiovascular disease (except hypertension controlled by medication);
* Physical impairments for exercise diagnosed through anamnesis;

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness evaluation change after 12 weeks | Testing of VO2peak change - Baseline and 12 week
  We created a protocol on the treadmill to determine the peak oxygen uptake change(VO2peak), the first ventilatory threshold and the second ventilatory threshold. The protocol consists in 1-minute stages. The initial speed is 1.86 miles per hour. In each stage, the speed increases 0.3 miles per hour and every 2 stages, the treadmill inclination increases 1%. The test is interrupted when the subject indicates exhaustion. The respiratory gases will be collected through a portable gas analyzer (VO2000, MedGraphics, Ann Arbor, USA).
  The maximum value of VO2 , closed to exhaustion will be considered the VO2peak. The fist and the second ventilatory threshold will be determined by the ventilation versus intensity curve and confirmed by the O2 and Carbon dioxide ventilatory equivalents by two independent physiologists in a visual inspection.

SECONDARY OUTCOMES:
Quality of Life change after 12 weeks (Score) | Baseline and 12 week
  World Health Organization Quality of Life-bref - WHOQOL-bref
Maximal dynamic strength change after 12 weeks (kg) | Baseline and 12 week
  maximum repetition of knee extensors
Maximal voluntary isometric contraction of knee extensors change after 12 weeks | Baseline and 12 week
  electromyography
muscle thickness of knee extensors change after 12 weeks | Baseline and 12 week
  ultrasound image
neuromuscular economy of vastus lateralis and rectus femoris change after 12 weeks | Baseline and 12 week
  electromyography
maximum muscular activity of vastus lateralis and rectus femoris change after 12 weeks | Baseline and 12 week
  electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Cristine Alberton, Phd, Principal Investigator — UFPel
Locations (1):
- Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul, Brazil